CLINICAL TRIAL: NCT00792272
Title: Prevalence of Aspirin Resistance in Hemodialysis Patients
Brief Title: Prevalence and Profile of Aspirin Resistance in Hemodialysis Patients
Status: Completed | Type: Observational
Sponsor: Northwell Health (Other)
Collaborators: Staten Island University Hospital (Other)
Responsible Party: Principal Investigator, Suzanne El-Sayegh, Assoc. Chair of Medicine, Northwell Health
Other Study IDs: 08-013
Record Dates: First submitted 2008-11-14; First posted 2008-11-17 (Estimated); Last update posted 2013-07-22 (Estimated); Status verified 2013-07

CONDITIONS: Aspirin Resistance
Keywords: aspirin resistance; aspirin resistance in hemodialysis patients

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Dialysis patient could be more aspirin resistant than the general population based on data from chronic kidney disease patients

DETAILED DESCRIPTION:
We will try to describe the profile of aspirin resistant patient in hemodialysis patients

ELIGIBILITY:
Inclusion Criteria:

* all hemodialysis patients on aspirin

Exclusion Criteria:

* low platelets <100.000
* coagulopathy, bleeding disorders
* patient on plavix

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all hemodialysis patients on aspirin
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2008-06; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Aspirin Resistance in Hemodialysis patients | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne El-Sayegh, MD, Principal Investigator — SIUH